CLINICAL TRIAL: NCT06243757
Title: Trans-Pacific Multicenter Collaborative Study of Minimally Invasive Proximal Versus Total Gastrectomy for Proximal Gastric and Gastroesophageal Junction Cancers
Brief Title: A Study of Minimally Invasive Proximal Gastrectomy Versus Minimally Invasive Total Gastrectomy for Gastric and Gastroesophageal Junction Cancers
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23-324
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Gastric Cancer; GastroEsophageal Cancer; Gastroesophageal Junction Adenocarcinoma
Keywords: gastric cancer; non-metastatic gastric cancer; Gastroesophageal Junction Adenocarcinoma; gastroesophageal cancer; GEJ adenocarcinoma; MIPG; MITG; Minimally Invasive Proximal Gastrectomy; Minimally Invasive total gastrectomy; 23-324; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Minimally Invasive Proximal Gastrectomy/MIPG: Participants will undergo MIPG (Trial Procedure)
  Interventions: Other: MDASI-GI
- Minimally Invasive Total Gastrectomy/MITG: Participants will undergo MITG (Standard of Care/Control Group)
  Interventions: Other: MDASI-GI

INTERVENTIONS:
Other: MDASI-GI — The MDASI-GI assesses 5 symptoms specific to gastrointestinal cancer:
  constipation diarrhea or watery stools difficulty swallowing change in taste feeling bloated
  Using this questionnaire, participants score the severity of their symptoms over the previous 24 hours on a scale of 0 (not present) to 10 (as bad as you can imagine).
  Other Names: MD Anderson Symptom Inventory for gastrointestinal cancer

SUMMARY:
Participants will a diagnosis of gastroesophageal junction (GEJ) adenocarcinoma and will have either a minimally invasive proximal gastrectomy (MIPG) or a minimally invasive total gastrectomy (MITG) as part of their routine care. Participants with complete a questionnaire 1 month before the surgical procedure and then 1, 3, 6 and 12 months after the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and read English, Spanish, Japanese or Korean
* Patients with a biopsy-confirmed diagnosis of non-metastatic gastric or GEJ adenocarcinoma, who are scheduled to undergo MIPG or MITG for curative-intention
* Age ≥ 18

Exclusion Criteria:

* Patients with known malabsorption syndromes or a lack of physical integrity of the upper gastrointestinal tract
* Patients with known narcotic dependence, with average daily dose > 5 mg oral morphine equivalent
* Subjects deemed unable to comply with study and/or follow-up procedures, at investigators' discretion
* Patients who are pregnant (since are excluded from receiving standard-of-care MIPG or MITG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The initial contact with the potential participants will be conducted either by the treatment team, investigator or the research staff working in consultation with the treatment team. Participants will be screened in gastric and mixed tumor surgery clinics on the 5th floor of the MSKCC 53rd Street outpatient clinic building. The investigator/research staff will review portions of the medical record to determine if they are eligible. Participants who are eligible will be approached by study personnel in clinic. The study will be explained to participants by the study personnel and interested participants will be given the consent form to review.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2036-01-08 (Estimated); Study Completion 2036-01-08 (Estimated)

PRIMARY OUTCOMES:
Appetite level score according to the MDASI-GI | 3 months after surgery
  The primary outcome is the appetite level score (with 0 being the best and 10 being the worst) according to the MDASi-GI at 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Strong, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York
  - MD Anderson Cancer Center (Data Analysis Only), Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org